CLINICAL TRIAL: NCT01239498
Title: Saline Injection - Assisted Anesthesia in Eyelid Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ido Didi Fabian MD, Sheba medical center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-8246-DF-CTIL
Record Dates: First submitted 2010-11-02; First posted 2010-11-11 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline + Lidocaine/Adrenaline (Experimental)
  Interventions: Procedure: Injection of Saline + Lidocaine/Adrenaline
- Lidocaine/Adrenaline only (Placebo Comparator)
  Interventions: Procedure: Lidocaine/Adrenaline only

INTERVENTIONS:
Procedure: Injection of Saline + Lidocaine/Adrenaline — All anaesthetic injections will consist of xylocaine 1% with 1:100,000 adrenaline and will be administered through a short 30 Gauge needle at a constant slow speed at multiple (6-7) sites along the upper lid by a single oculoplastic consultant.
  The experimental eyelid will receive a saline-consisted injection 0.5cc prior to the administration of the anesthetic injection.
  Injection of Saline + Lidocaine 1%
  Other Names: Local eyelid anesthesia
  Arms: Saline + Lidocaine/Adrenaline
Procedure: Lidocaine/Adrenaline only — Injection of Lidocaine/Adrenaline only
  Other Names: Local eyelid anesthesia
  Arms: Lidocaine/Adrenaline only

SUMMARY:
The investigators hypothesize that injection of saline to the upper eyelids prior to lidocaine/adrenaline injection will reduce pain of the local anesthetic in comparison to injection of lidocaine alone.

DETAILED DESCRIPTION:
Purpose:

To carry out a prospective randomised controlled clinical trial to compare the efficacy of saline injection prior to the injection of Lidocaine/Adrenaline in reducing the pain of local anaesthetic injections into the upper eyelid.

Hypothesis:

Injection of saline to the upper eyelids prior to lidocaine/adrenaline injection reduces the pain of anaesthetic injections in upper eyelid surgery.

Justification:

In many surgical procedures performed under local anaesthetic, the most frightening and painful aspect of the procedure for patients is the anaesthetic injection, and various techniques have been advocated to address this.

Simple measures that reduce the pain of anaesthetic injection and are widely practised include administering the injection slowly and using a fine-bore needle (30 Gauge). Other techniques that have been shown to be effective include warming or buffering the local anaesthetic. The use of 0.9% bacteriostatic saline solution in conjunction with lidocaine has been demonstrated to significantly reduce patients' perceived pain during the injection and operative procedure in eyelid surgery. Cooling the skin immediately prior to treatment has been shown to reduce the pain of dermatological laser procedures although this might be difficult to perform around the eyes because of the risk of injuring the cornea. Similarly, topical anaesthetic agents, such as EMLA (eutectic mixture of local anaesthetics) cream, which are applied to the skin one hour prior to injection are commonly employed for use on the limbs of infants and children but are not safe for use around the eyes since inadvertent ocular application causes corneal de-epithelisation.

Sedative agents, such as midazolam may be useful in anxious patients, but this requires the input of an anaesthetist and it is often difficult to finely control the level of sedation; it is usually preferable not to have patients sedated during eyelid surgery when patient cooperation is required intra-operatively to assess the height of the eyelids, for example in ptosis surgery.

The investigators have noticed in clinical practice that whenever the investigators injected saline into the upper eyelids prior to the injection of the mixture of lidocaine/adrenaline the patients reported of no pain. The investigators assume that by using the isotonic saline cells in the tissue are not harmed and a minor effect of anesthesia is achieved. The anesthetic solution injected later on is diluted, however the eyelid is properly anesthesized.

Research Methods:

The study will be a prospective, interventional, randomised, controlled clinical trial.

All patients who fit the inclusion criteria will be offered participation in the trial on the day their surgery is booked. They will be given an information leaflet about the trial, explaining the aim of the study without describing the effect of the saline injection prior to the anesthetic solution injection in order to reduce the risk of biasing their perception. They will be advised that non-participation will not affect their care in anyway.

The intervention is of no risk to the patient and will not affect the surgical procedure in any way. Any questions that the patient has will be addressed beforehand and they will be required to sign a consent form prior to inclusion in the trial.

They will be advised beforehand that they will be required to verbally rate their pain score on a scale of 0 to 10 immediately after both sides have been anaesthetised, with 0 being no pain and 10 being the worst imaginable pain.

All participants included in the study will undergo bilateral surgery and will therefore act as their own controls: Saline will only be injected prior to the injection of the anaesthetic into one side. The test and placebo will be randomly assigned to either the first or second eyelid; the right eyelid will be injected first in all patients, as is routine practice. Computer-generated sequential binary randomisation will be used. Allocation will be concealed from the surgeon until immediately prior to the anaesthetic injection.

All anaesthetic injections will consist of xylocaine 1% with 1:100,000 adrenaline and will be administered through a short 30 Gauge needle at a constant slow speed at multiple (6-7) sites along the upper lid by a single oculoplastic consultant.

Patients' verbal pain scores will be elicited and documented immediately by the oculoplastic fellow.

Planned sample size On a scale of 0 to 10 a difference in pain score of 1.5 may be considered to be clinically significant. The power calculation for a paired t-test with 90% power and p=0.05 demonstrated that a sample size of 80 patients to be more than sufficient to detect a significant difference.

The results will be submitted for publication in a peer-reviewed ophthalmological journal and presentation at international ophthalmological meetings.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing bilateral upper eyelid surgery under local anaesthetic who have given fully informed consent to be in the trial

Exclusion Criteria:

* Previous upper eyelid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Patients' verbal pain scores will be elicited and documented immediately by the oculoplastic fellow | 1-2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ido Didi Fabian, MD, Study Chair — Sheba medical center, Goldschleger institute
Locations (2):
- Israel (2):
  - Goldschlager eye institute, Ramat Gan
  - Goldschleger institute of ophthalmology, Sheba medical center, Ramat Gan

REFERENCES:
- [Background] Chen BK, Eichenfield LF. Pediatric anesthesia in dermatologic surgery: when hand-holding is not enough. Dermatol Surg. 2001 Dec;27(12):1010-8. doi: 10.1046/j.1524-4725.2001.01854.x. PMID 11849262
- [Background] Brogan GX Jr, Giarrusso E, Hollander JE, Cassara G, Maranga MC, Thode HC. Comparison of plain, warmed, and buffered lidocaine for anesthesia of traumatic wounds. Ann Emerg Med. 1995 Aug;26(2):121-5. doi: 10.1016/s0196-0644(95)70139-7. PMID 7618771
- [Background] Bainbridge LC. Comparison of room temperature and body temperature local anaesthetic solutions. Br J Plast Surg. 1991 Feb-Mar;44(2):147-8. doi: 10.1016/0007-1226(91)90050-t. PMID 2018901
- [Background] Stewart JH, Cole GW, Klein JA. Neutralized lidocaine with epinephrine for local anesthesia. J Dermatol Surg Oncol. 1989 Oct;15(10):1081-3. doi: 10.1111/j.1524-4725.1989.tb03127.x. PMID 2794204
- [Background] Bartfield JM, Gennis P, Barbera J, Breuer B, Gallagher EJ. Buffered versus plain lidocaine as a local anesthetic for simple laceration repair. Ann Emerg Med. 1990 Dec;19(12):1387-9. doi: 10.1016/s0196-0644(05)82603-4. PMID 2240750
- [Background] Fayers T, Morris DS, Dolman PJ. Vibration-assisted anesthesia in eyelid surgery. Ophthalmology. 2010 Jul;117(7):1453-7. doi: 10.1016/j.ophtha.2009.11.025. Epub 2010 Mar 19. PMID 20303597